CLINICAL TRIAL: NCT03602963
Title: A Comparative Study on the Accuracy and Usability Between the Dexcom G5 Mobile CGM System and the FreeStyle Flash Glucose Monitoring System
Brief Title: Comparison Between Dexcom G5 Mobile Continuous Glucose Monitoring (CGM) System and the FreeStyle Libre Flash Glucose Monitoring System
Status: Completed | Type: Observational
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: JessaH_18.64/ped18.02
Record Dates: First submitted 2018-07-05; First posted 2018-07-27 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2018-07

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes Mellitus; Child; Glucose sensor; Accuracy; Usability
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Dexcom G5 mobile CGM system: Children (6 to 18 years) with type 1 diabetes mellitus treated with insulin injections and wearing a FreeStyle Libre Flash glucose sensor that will switch to the Dexcom G5 mobile glucose monitoring system.
  Interventions: Device: Dexcom G5 Mobile CGM system

INTERVENTIONS:
Device: Dexcom G5 Mobile CGM system — The accuracy and usability ot the Dexcom G5 mobile CGM system will be evaluated

SUMMARY:
1. The accuracy of the sensors (Dexcom G5 vs FreeStyle Libre Flash glucose monitoring) will be evaluated by simultaneous wearing of the 2 sensors during 2 weeks. During these 2 weeks the patients will do at least four capillary blood glucose measurements to compare with the sensor results.
2. Patient satisfaction will be evaluated using a questionnaire that will be completed after the Dexcom G5 sensor has been worn for 1 month.
3. The data recorded by the FreeStyle Libre Flash glucose monitoring system (average glucose,% above target, % within target, % under target, amount of hypoglycemia) in the month prior to the 2 weeks of double sensor wear will be compared to the same data recorded by the Dexcom G5 mobile CGM system during the first month of use.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus
* Treated by insulin injections

Exclusion Criteria:

* Other types of diabetes
* Treated with insulin pump

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with type 1 diabetes mellitus treated with insulin injections
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Accuracy of the Dexcom G5 mobile continuous glucose monitoring (CGM) system by comparison of sensor glucose measurements with capillary blood glucose determinations | 2 weeks
  Comparison of sensor glucose measurements will be compared with capillary blood glucose measurements at least 4 times a day

SECONDARY OUTCOMES:
Patients' and parents' satisfaction with the Dexcom G5 mobile CGM system will be evaluated by a standardized questionnaire | 1 month
  Patients' and parents' satisfaction with the Dexcom G5 mobile CGM system will be evaluated by a standardized questionnaire after 1 month of sensor wear. Patients and parents will rate their experience with the Dexcom G5 mobile CGM system on a scale of 1 (strongly agree) to 5 (strongly disagree). There are three questions about sensor application (e.g. It is easy to put the sensor on) and eleven questions about the wearing of the sensor (e.g. The sensor doesn't disturb me for sporting).

CONTACTS AND LOCATIONS:
Overall Officials: Guy Massa, MD, PhD, Principal Investigator — Jessa Hospital
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Undecided